CLINICAL TRIAL: NCT00187655
Title: Effect of Genetic Variation in the Transporter, OAT3, on the Renal Secretion of Cefotaxime
Brief Title: Effect of, OAT3, on the Renal Secretion of Cefotaxime
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 867
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2014-05-12 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Focus Groups
Keywords: Healthy volunteers willing to be dosed with cefotaxime
MeSH Terms: interventions — Cefotaxime

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cefotaxime (Other): Cefotaxime will be administered as a single IV push of 2 grams over 5 minutes.
  Interventions: Drug: Cefotaxime

INTERVENTIONS:
Drug: Cefotaxime — Cefotaxime will be administered as a single IV push of 2 grams over 5 minutes.
  Other Names: Claforan; Cefotaxime Sodium

SUMMARY:
In the proposed study, we plan to use a genotype to phenotype strategy to study the role of the organic anion transporter, OAT3, in drug response. More specifically we will examine the contribution of OAT3 to the renal clearance of anionic drugs such as cefotaxime by studying individuals with a non-functional (or poorly-functional) variant of OAT3.

DETAILED DESCRIPTION:
Traditionally, clinical pharmacogenetic studies have begun with identifying a known phenotype (e.g., an aberrant response to a drug) followed by isolating the variant protein and gene responsible for that phenotype. With the sequence of most human genes known, it is possible to carry out pharmacogenetic studies in the reverse manner (i.e., genotype to phenotype). Patients with a known variant of a gene can be studied for their response to certain drugs, which can help elucidate the importance of that gene in drug response. In the proposed study, we plan to use a genotype to phenotype strategy to study the role of OAT3 and related variants in drug response.

Renal elimination of anionic drugs occurs by filtration and active secretion. For secretion, the drug is transported from the blood into the renal tubular cell through the basolateral membrane. This transport occurs against both a concentration and electrochemical gradient, and must therefore be mediated by organic anion transporters (OATs). To date, six human OATs have been identified, OAT 1-5, and OAT7. OAT1 and OAT3 are the dominant OATs found on the basolateral aspect of the renal proximal tubular cells and are hence suspected of playing a significant role in renal anionic drug elimination [3, 4].

Active renal tubular secretion of most beta-lactam antibiotics, including cephalosporins, has long been recognized, with OATs likely playing a major role, though the relative role of each is unclear [5]. In vivo studies have demonstrated that the cephalosporin cefotaxime has a ten-fold higher affinity for OAT3 than OAT1 [6]. Thus, patients with OAT3 variants would be expected to exhibit altered renal secretion of cefotaxime.

Cefotaxime is a common cephalosporin used in the treatment of bacterial infections. Dosed up to 1-2 mg every 6-8 hours, it has been shown to be safe in patients with normal renal function. Cefotaxime is given intravenously, and is metabolized to desacetyl cefotaxime (DACM) which retains antibacterial activity. DACM is further metabolized to two inactive metabolites, M2 and M3; all four forms of cefotaxime are renally eliminated, with active secretion representing a significant percentage of total clearance (44% for cefotaxime, 64% for DACM) [7]. The half-life of cefotaxime and DACM are 1 and 1.5 hours, respectively. Patients with poorly functional OAT3 and related variants might be expected to exhibit reduced tubular secretion of both cefotaxime and its metabolites, and result in higher or prolonged blood levels. Because such variants may reduce the amount of cefotaxime that enters the tubular cells, they may also be associated with a reduced incidence of cephalosporin-induced nephrotoxicity.

The PMT group has a collection of 500 DNA samples from young, healthy adults from four major ethnic groups (125 each from Caucasians, African-Americans, Mexicans, and Chinese). This collection (The Pharmacogenetics of Membrane Transporters), is referred to as "SOPHIE" (Study of Pharmacogenetics in Ethnically-diverse Populations), and includes only volunteers who have consented to be called back for consideration of enrollment in future studies.

In recent studies, we identified nine non-synonymous OAT3 variants among subjects participating in the SOPHIE study. We cloned and introduced each variant into a heterologous expression system and tested the encoded transporters for their ability to transport estrone sulfate (a documented substrate for OAT3). Four variants were identified that resulted in a complete loss of function: F129L (in one Hispanic subject), R149S (in an Caucasian and an African American subject), Q239stop (in the same African American subject), and R277W (in an Asian subject). In the subject with two non-functional variants, it is unknown whether the variants occur on the same chromosome, or if the variants are on different chromosomes. The latter would potentially make the subject completely OAT3 deficient. An additional variant (I305F) which showed reduced transport ability for some, but not all, OAT3 substrates was identified in three Asian and one Hispanic subject. One variant (A310V) which showed increased transport of estrone sulfate compared to the common allele was identified in a single Caucasian subject.

This study will address the following question: Do individuals who carry altered-function in OAT3 and related variants exhibit differences in the pharmacokinetics of cefotaxime in comparison to individuals who carry the common allele?

ELIGIBILITY:
Inclusion Criteria:

1. Previous participation in the "SOPHIE" study;
2. Has a specific genotype for OAT3

Exclusion Criteria:

1. Under 18 years old or over 45 years old;
2. Pregnant (pregnancy status in female subjects will be determined by a urine pregnancy test before study drug administration);
3. They report a prior history of any allergic reaction to cephalosporin antibiotic, or severe hypersensitivity to penicillin;
4. Has a prior history of renal or hepatic dysfunction (renal and hepatic function will also be determined for each subject with prescreening blood tests);
5. Taking a medication that could confound study results (such as known substrates or inhibitors of OATs);
6. They do not consent to participate in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2004-01; Primary Completion 2011-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Giacomini, PhD, Principal Investigator — University of California, San Francisco

REFERENCES:
- [Result] Erdman AR, Mangravite LM, Urban TJ, Lagpacan LL, Castro RA, de la Cruz M, Chan W, Huang CC, Johns SJ, Kawamoto M, Stryke D, Taylor TR, Carlson EJ, Ferrin TE, Brett CM, Burchard EG, Giacomini KM. The human organic anion transporter 3 (OAT3; SLC22A8): genetic variation and functional genomics. Am J Physiol Renal Physiol. 2006 Apr;290(4):F905-12. doi: 10.1152/ajprenal.00272.2005. Epub 2005 Nov 15. PMID 16291576

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment concluded with 24 subjects and study is in analysis phase. Recruitment of subjects were At the CRC at SFGH. Dates of recruitment 2004-9/2011.
Pre-assignment Details: No wash-out as these were healthy control subjects not currently on any medications.
Period: Overall Study
Arm/Group | Cefotaxime
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cefotaxime
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Effect of OAT3 on Renal Secretion of Cefotaxime IV Based on Genotype
Description: Participants were stratified by their OCT3 genotype, heterozygous vs homozygous. The renal clearance of cefotaxime was measured by urine content of cefotaxime metabolites in participants after the single IV push administration of 2 grams of cefotaxime.
Time Frame: post dose up to 24 hours
Population: The OAT3 Ile305Phe variant was determined to be heterozygous or homozygous for each healthy participant.
Measure: Mean (Standard Deviation); unit: mL/min
Groups:
- Heterozygous for the Ile305Phe Variant: 2 grams of Cefotaxime was administered as a single IV push of 2 grams over 5 minutes into healthy individuals that were identified as heterozygous for the Ile305Phe variant and compared to volunteers that were homozygous for the reference allele. Renal clearance and net secretory component of cefotaxime renal clearance (CLsec ) were analyzed.
- Homozygous for OAT3-Ile305Phe Variant: 2 grams of Cefotaxime was administered as a single IV push of 2 grams over 5 minutes into healthy individuals that were identified as homozygous for the Ile305Phe variant and compared to volunteers that were heterozygous for the reference allele. Renal clearance and net secretory component of cefotaxime renal clearance (CLsec ) were analyzed.
Arm/Group | Heterozygous for the Ile305Phe Variant | Homozygous for OAT3-Ile305Phe Variant
Number analyzed (Participants) | 12 | 12
mL/min | 84.8 (32.1) | 158 (44.1)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from 2004-2011 or enrollment period of study.
Description: No Adverse events were reported throughout the study.
Arm/Group | Cefotaxime
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes